CLINICAL TRIAL: NCT05672264
Title: Whole-body Electromyostimulation for the Treatment of Knee Osteoarthritis (EMSOAT) in Overweight People - a Randomized Controlled Trial
Brief Title: Whole-Body Electromyostimulation and Knee Osteoarthritis
Acronym: EMSOAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKER_EMS_Knee
Record Dates: First submitted 2023-01-02; First posted 2023-01-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WB-EMS group (Experimental): WB-EMS application
  Interventions: Other: Whole-Body Electromyostimulation
- Control (Active Comparator): Standardised physiotherapy (six sessions)
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Whole-Body Electromyostimulation — Consistently supervised, video-guided WB-EMS application 1.5 times per week for 28 weeks. Bipolar electric current with a frequency of 85Hz, an impulse-width of 350 µs will be used in an interval approach with 6 sec of EMS stimulation with a direct impulse boost and 4 sec of rest. Low intensity movements or exercises in a standing position were performed during the 6 s stimulation period.
  Arms: WB-EMS group
Other: Physiotherapy — Six standardised physiotherapy sessions (20 min each)
  Arms: Control

SUMMARY:
The aim of the present study is to evaluate the effects of WB-EMS application in overweight women and men with knee osteoarthritis, with special consideration of sustainability. In this randomised controlled trial 72 overweight patients with knee osteoarthritis aged 40-70 years will be included and randomly assigned to two groups (WB-EMS vs. control group (CG)). The intervention group will perform six WB-EMS sessions/month of 20 min for 6 months. An intermittent low frequency WB-EMS-protocol with an impulse phase of 6s, followed by an impulse break of 4s will be applied. The control group will undergo a tailored physiotherapy program of 6 sessions defined as usual care. In addition, both groups will complete a self-management training programme for osteoarthritis of 6 sessions over 12 weeks.

DETAILED DESCRIPTION:
Studies consistently show a positive effect of strength training on pain and function in knee osteoarthritis. In addition to local neuromuscular effects, systemic mechanisms that modulate inflammatory processes are increasingly being discussed as mechanisms of action. Overweight and obesity might be involved in this process. Despite high evidence, unfortunately only few people with osteoarthritic knee pain are willing or able to perform conventional muscular strength training on a regular basis. In this context, whole-body electromyostimulation (WB-EMS) is a time-efficient, joint-friendly and subjectively less strenuous training alternative. In WB-EMS, all large muscle groups of the body are simultaneously activated and brought to contraction by electrical impulses. Together with easy movements with minor mechanical stress on the knee joint, the additive WB-EMS activates muscle contraction and results in measurable muscular effects.

The aim of the present study is to evaluate the effects of a 6-month WB-EMS application in overweight women and men with knee osteoarthritis, with special consideration of sustainability. In this randomised controlled trial (RCT) 72 overweight patients (BMI >25 kg/m2) with knee osteoarthritis (radiographic severity Kellgren-Lawrence 2 and 3) aged 40-70 years will be included and randomly assigned to two groups (WB-EMS vs. control group (CG)). The intervention group will perform six WB-EMS sessions/month of 20 min for 6 months. An intermittent low frequency WB-EMS-protocol (85 Hz, 350 µs) with an impulse phase of 6s, followed by an impulse break of 4s will be applied. The control group will undergo a tailored physiotherapy program of 6 sessions defined as usual care. In addition, both groups will complete a self-management training programme for osteoarthritis of 6 sessions over 12 weeks.

At baseline, after 6 months of intervention and after a further 6 months of follow-up, knee pain and function will be determined by the KOOS instrument (Knee Injury and Osteoarthritis Outcome Score). Functional tests and isokinetic leg strength measurements will also be performed. In parallel, MRI assessments are applied to quantify effects on joint structure (whole organ assessment; MRI Osteoarthritis Knee Score (MOAKS)) and visceral fat as well as muscle quality changes at the mid-thigh. Whole body composition analyses are performed using segmental whole-body bioimpedance analysis (BIA) for quantification of body fat and fat-free mass. Blood samples are obtained at baseline, 6 and 12 months to determine inflammatory biomarkers (CRP, IL-1beta, MMP-3) and cartilage formation (PIINP).

The study will provide evidence and detailed insights of the WB-EMS induced effects on pain, function, muscle structure and strength, body composition, joint tissues and anti-inflammatory effects in knees with osteoarthritis. From a clinical perspective, the study will provide important information regarding a promising non-pharmacological therapeutic approach for the treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* overweight (BMI>25 kg/m2)
* radiographically confirmed early to moderate femorotibial osteoarthritis (Kellgren- Lawrence grades 2 and 3)
* osteoarthritic knee pain for at least 3 months
* average pain intensity > 2.5 (NRS 0-10)

Exclusion Criteria:

* WB-EMS in the last year or resistance exercise >1 session/week in the last year
* present glucocorticoid or opioid medication
* trauma of the knee joint within the last 3 months
* intra-articular injections in the knee joint within the last 3 months
* malignant diseases
* serious cardiovascular diseases
* conditions or diseases that are contraindications for WB-EMS
* absence ≥3 weeks during the intervention period

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Knee pain | baseline to 6 month follow up
  Changes in pain of the knee joint as determined by the Knee Injury and Osteoarthritis Outcome Score (KOOS) in the WB-EMS- compared to changes in the control group.KOOS score for "knee pain" vary from 1 (never/no pain) to 5 (always/very severe pain)

SECONDARY OUTCOMES:
Self rated symptoms | baseline to 6-month follow-up
  Changes in Knee Injury and Osteoarthritis Outcome Score (KOOS)-dimension "self-rated symptoms" in the WB-EMS- compared to changes in the control group. KOOS score for "self related symptoms" vary from 1 (never) to 5 (always).
Knee stiffness | baseline to 6-month follow-up
  Changes in Knee Injury and Osteoarthritis Outcome Score (KOOS)-dimension "knee stiffness" in the WB-EMS- compared to changes in the control group. KOOS score for "knee stiffness" vary from 1 (no problems) to 5 (very hard).
Function in daily living | baseline to 6-month follow-up
  Changes in Knee Injury and Osteoarthritis Outcome Score (KOOS)-dimension "function in daily living" in the WB-EMS- compared to changes in the control group. KOOS score for "function in daily living" vary from 1 (no problems) to 5 (very serious problems).
Function in sports and recreational activities | baseline to 6-month follow-up
  Changes in Knee Injury and Osteoarthritis Outcome Score Knee Injury and Osteoarthritis Outcome Score (KOOS)-dimension "function in sports and recreational activities" in the WB-EMS- compared to changes in the control group. KOOS score for "function in sports and recreational activities" vary from 1 (no problems) to 5 (very serious problems).
Quality of Life | baseline to 6-month follow-up
  Changes in Knee Injury and Osteoarthritis Outcome Score (KOOS)-dimension "quality of life" in the WB-EMS- compared to changes in the control group. KOOS score for "quality of life vary" from 1 (never/no problems) to 5 (always/very serious problems).
Total Knee Injury and Osteoarthritis Outcome Score (KOOS) score | baseline to 6-month follow-up
  Changes in total KOOS-score in the WB-EMS- compared to changes in the control group. Average total KOOS score vary" from 1 (never/no problems) to 5 (always/very serious problems).
Pain intensity of the knee | baseline to 6-month follow-up
  Changes in pain intensity of the knee as determined by a 7-day knee pain protocol (applying the NRS 0-10 scale) in the WB-EMS- compared to changes in the control group.
Joint and cartilage structure | baseline to 6-month follow-up
  Changes in joint and cartilage structure as determined by the MRI Osteoarthritis Knee Score (MOAKS) in the WB-EMS- compared to changes in the control group.
Intrafascial muscle tissue at the mid-thigh | baseline to 6-month follow-up
  Changes in volume adjusted intrafascial muscle tissue volume (MT) at the mid-thigh, as determined by MRI in the WB-EMS- compared to changes in the control group.
Intermuscular adipose tissue at the mid-thigh | baseline to 6-month follow-up
  Changes in volume adjusted intermuscular adipose tissue (IMAT) at the mid-thigh, as determined by MRI in the WB-EMS- compared to changes in the control group.
Intrafascial fat fraction at the mid-thigh | baseline to 6-month follow-up
  Changes in volume adjusted intrafascial fat fraction (IFFF) at the mid-thigh, as determined by MRI in the WB-EMS- compared to changes in the control group.
Visceral fat mass | baseline to 6-month follow-up
  Changes in visceral fat mass as determined by determined by MRI in the WB-EMS- compared to changes in the control group.
C-reactive Protein (CRP) | baseline to 6-month follow-up
  Changes in CRP-levels in the WB-EMS- compared to changes in the control group.
Interleukin 1beta (IL1beta) | baseline to 6-month follow-up
  Changes in IL1beta-levels in the WB-EMS- compared to changes in the control group.
Matrix metalloprotease 3 (MMP-3) | baseline to 6-month follow-up
  Changes in MMP-3 levels in the WB-EMS- compared to changes in the control group.
Serum N-terminal pro-peptide of collagen IIA (PIINP) | baseline to 6-month follow-up
  Changes in PIINP levels in the WB-EMS- compared to changes in the control group.
Maximum strength of the hip-/leg extensors | baseline to 6-month follow-up
  Changes in maximum strength of the hip-/leg extensors as determined by an isokinetic leg press in the WB-EMS- compared to changes in the control group.
Chair Rise Test | baseline to 6-month follow-up
  Changes in the 30-second Chair Rise Test in the WB-EMS- compared to changes in the control group.

OTHER OUTCOMES:
Drop-out rate | baseline to 6-month follow-up
  Drop-out rate of the WB-EMS- compared to the control group.
Attendance rate | baseline to 6-month follow-up
  Attendance rate in the WB-EMS group (in percent of maximum sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Kast, MSc, Principal Investigator — Institute of Radiology, University Hospital-Nürnberg
Locations (1):
- Institute of Medical Physics University of Erlangen-Nurnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kemmler W, Kleinoder H, Frohlich M. Editorial: Whole-body electromyostimulation: A training technology to improve health and performance in humans? volume II. Front Physiol. 2022 Aug 5;13:972011. doi: 10.3389/fphys.2022.972011. eCollection 2022. No abstract available. PMID 36111142
- [Result] Bloeckl J, Raps S, Weineck M, Kob R, Bertsch T, Kemmler W, Schoene D. Feasibility and Safety of Whole-Body Electromyostimulation in Frail Older People-A Pilot Trial. Front Physiol. 2022 Jun 24;13:856681. doi: 10.3389/fphys.2022.856681. eCollection 2022. PMID 35812334
- [Result] Kemmler W, Shojaa M, Steele J, Berger J, Frohlich M, Schoene D, von Stengel S, Kleinoder H, Kohl M. Efficacy of Whole-Body Electromyostimulation (WB-EMS) on Body Composition and Muscle Strength in Non-athletic Adults. A Systematic Review and Meta-Analysis. Front Physiol. 2021 Feb 26;12:640657. doi: 10.3389/fphys.2021.640657. eCollection 2021. PMID 33716787